CLINICAL TRIAL: NCT03815227
Title: Outpatient Birth: Pilot Study to Assess the Feasibility of Maternity Out the Same Date or the Next Day of the Birth
Brief Title: Outpatient Birth: Pilot Study
Acronym: ACCAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-06-CHRMT
Record Dates: First submitted 2019-01-23; First posted 2019-01-24 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Outpatient Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outpatient birth (Experimental): Maternity out the same date or the next day of the birth
  Interventions: Other: Outpatient birth

INTERVENTIONS:
Other: Outpatient birth — Maternity out the same date or the next day of the birth and home-based follow up with a liberal midwife

SUMMARY:
The diminution of the average length stay (ALS) in French maternity is a clear evolution, the objective of the draft law on social security is to reduce the ALS to equal other OECD countries. The over-medicalization of maternal health raises the question of relevant and iatrogeny of Professional practices. Furthermore, pregnant woman, future parents expressed their wish for an individual support and more physiological respectful. A more-effective Professional coordination is expected where the midwife is a major player.

DETAILED DESCRIPTION:
The aim of the study is to identify and evaluate an outpatient birth path during the first 24 hours after the birth.

ELIGIBILITY:
Inclusion Criteria:

* With no multiple pregnancy, of less than 20 weeks of gestation
* With a BMI between 17,5 and 35 kg/m²
* is able to understand research's informations
* affiliated member of the social security system
* Have given an informed consent

Exclusion Criteria:

* With psychological vulnerability, social vulnerability, addictions and high dependency
* With an unbalanced chronic pathology or susceptible to contraindicated a physiologic birth
* With history of caesarean, foeto-maternal incompatibility, gestational hypertension, pre-eclampsia, HELLP syndrome or retro-placental hematoma, sphincter tear
* With history of birth with perinatal asphyxia and sequelae or an unexplained perinatal death
* With history of puerperal psychosis
* Under guardianship

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant woman
Enrollment: 50 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Output rate | Day 1
  Output rate within 24 hours of birth

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Thionville, Moselle, France